CLINICAL TRIAL: NCT04140617
Title: Bystanders' Exposure to Electronic Cigarette Aerosol in Confined Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Català d'Oncologia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TackSHS WP8 Experimental
Record Dates: First submitted 2019-10-01; First posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Secondhand Exposure to Electronic Cigarette
Keywords: vaping; electronic cigarette; passive exposure; e-cigarette
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-cigarette aerosol exposure in a room (Experimental): Exposure to aerosol of electronic cigarette produced by experienced user (30 minutes of exposure) in a 25 m3 room.
  Interventions: Behavioral: Exposure to aerosol of electronic cigarette
- E-cigarette aerosol exposure in a car (Experimental): Exposure to aerosol of electronic cigarette produced by experienced user (30 minutes of exposure) in a car.
  Interventions: Behavioral: Exposure to aerosol of electronic cigarette

INTERVENTIONS:
Behavioral: Exposure to aerosol of electronic cigarette — Exposure to aerosol of electronic cigarette (30 min)

SUMMARY:
Objective of this study is to investigate the bystanders' exposure to e-cigarette emissions in controlled conditions in confined settings.

Design: a cross-sectional experimental study developed in two settings: a car and a room. The experimental study will be replicated 5 times in each setting.

Three volunteers will be enrolled: 2 non-users of e-cigarettes (and non-smokers of any tobacco or nicotine product) and 1 exclusive e-cigarette user (not using any other tobacco or nicotine product) to create aerosol.

In brief, during the experimental session the e-cigarette user will be asked to use electronic cigarette during 30 minutes and two non-smokers will sit next to the user.

Individual exposure will be measured through saliva sample collection and irritation symptoms questionnaire to be collected 4 times: before exposure, just after 30 minutes of exposure, 30 minutes after the end of exposure and 3 hours after the end of exposure. Moreover, environmental exposure will be measured prior (5 min), during (30 min) and after (5 min) the exposure; particulate matter and airborne nicotine concentrations will be measure for this purpose.

DETAILED DESCRIPTION:
Objective: to investigate the bystanders' exposure to e-cigarette emissions in controlled conditions in confined settings.

Methods

Study design: this is a cross-sectional experimental study developed in two settings: a car and a room. The experimental study will be replicated 5 times in each setting.

It is important to notice that this study is an ad hoc experiment with volunteers and therefore it is not a clinical trial.

Study population: 3 volunteers will be enrolled: 2 non-users of e-cigarettes (and non-smokers of any tobacco or nicotine product) and 1 exclusive e-cigarette user (not using any other tobacco or nicotine product). Participants will be recruited through personal contacts of the research team and, if necessary, through social networks. All volunteers will receive a compensation for their participation in all replicates in both settings.

Thus, the participation of three volunteers will be required:

1. Two healthy non-smokers, one male and one female, to be exposed to e-cigarette emissions
2. One healthy e-cigarette user, to create the e-cigarette exposure

Each volunteer will be given appropriate information about the experiment, including its potential health effects.

Experiment Conditions

In order to investigate the passive exposure to the aerosol produced by e-cigarette use in healthy volunteers in controlled conditions, the following procedures will be performed:

* One week prior to the experiments a briefing session will be conducted inviting all three participants to provide them detailed information about the study and to explain the process of the experiment. During this day the information sheet will be provided to the participants and those willing to participate will sign a written consent form.
* Similar-to-real-life exposure to e-cigarette aerosol will be emulated by the use of one e-cigarette in each of the confined spaces.
* The experiment will be done in conditions with a relative humidity lower than 85% to obtain reliable measurements of airborne markers.
* Any system of ventilation, heating or air conditioning during the experiment will be avoided.
* During different periods of time, environmental and biological samples will be collected to objectively measure passive exposure to aerosol produced by the use of the e-cigarette.
* Some observational information regarding the environmental conditions, e-cigarette use and potential short-term health effects will be also gathered during the experiment.
* The experiment will be replicated in 5 consecutive days in each setting, from Monday to Friday. After each daily replication, the setting will be ventilated and will be only used for the following replication.
* First conduct the experiment in the car will be conducted and after at least 10 days the experiment in the room will be performed, to assure no biological exposure will remain in the bodies of non-smoker participants.

Particular conditions in the car

A similar-to-real-life exposure to e-cigarette aerosol will be emulated in a medium-size car by the use of one e-cigarette.

* The experiment will include a driver, 1 e-cigarette user, 2 non-smokers and a researcher.
* All the procedures will last 40 minutes:

  1. 5 minutes of baseline environmental and biological measurements. During this period the car will be stopped.
  2. 30 minutes of exposure to aerosol produced by an e-cigarette: the e-cigarette user will be asked to use the e-cigarette ad libitum. During this period, environmental measurements will be done and observational data will be collected. The car will be running continuously on a short circuit of 1.3 km at a speed of up to 70 km/h, with the front windows semi-open and the rear windows closed. During this period the car will be moving.
  3. 5 minutes of environmental measurement as an indicator of residual exposure. A biological measurement will be also done during these 5 mins. During this period the car will be stopped.

Particular conditions in the room

A similar-to-real-life exposure to e-cigarette aerosol will be emulated in a room of about 20-30 m3 by the use of one e-cigarette.

* The experiment will include 1 e-cigarette user, 2 non-smokers and a researcher, who will be seated around a table.
* All the procedures will last 40 minutes:

  1. 5 minutes of baseline environmental and biological measurements.
  2. 30 minutes of exposure to aerosol produced by an e-cigarette: the e-cigarette user will be asked to use the e-cigarette ad libitum. During this period, environmental measurements will be done and observational data will be collected.
  3. 5 minutes of environmental measurement as an indicator of residual exposure. A biological measurement will be also done during these 5 mins.

After the experiments

Once the experiments are finished, the participants will move to a different room and they will remain there for additional 3 hours. It will not be allowed to use e-cigarette during that period of time.

Biological measurements will be taken from all participants at 30 minutes and at 3 hours after finishing the experiment.

Measurements

Environmental measurements

Airborne nicotine. Nicotine will be collected using a sampler device of 37 mm in diameter containing a filter treated with sodium bisulphate. The sampler device will be connected to an air pump (flow 3 L/min) for active measurement. Two nicotine monitors will be used during the experiments in the car and two during the experiment in the room.

Particulate matter: Real-time measurement of airborne PM2.5 concentration will be done with a TSI SidePak AM510 at 1-sec interval and 10-min interval, respectively. Data will be downloaded to a local computer from internal storage for further data analyses.

Biological measurements

Saliva sample: Saliva samples will be collected from all participants four times in each experiment session: while measuring baseline environmental measurements, just at the end of the proper experiment period (exposure times), after 30 min and after 3 h of the exposure period. Saliva samples will be prepared into 2 aliquots for storage at -20 Cº at ICO. At the end of all the experiments saliva samples will be analysed to determine the concentration of nicotine and its main metabolites such as cotinine, 3'-OH-cotinine and nornicotine (in nl/mL), tobacco-specific nitrosamines (NNN, NNK and NNAL, in pg/mL), propylene glycol and glycerol (in nmol/mL).

Data Management

All data from questionnaires, environmental measurements and saliva analysis will be managed by researchers from the Tobacco Control Unit (UCT) at the Catalan Institute of Oncology (ICO).

Data will be collected in paper and will be digitalised in a protected database. All the samples will have a unique code to be linked with the already anonymised data from the questionnaires, and this data will be stored in the same database. Only a selected number of pre-designated members of the research team (who will sign a confidentiality document) will have access to the database and the freezer with the biological samples.

Selected personal data, including the names of respondents, will be collected separately to enable quality assurance procedures and to allow participants' willingness to withdraw from participation in the study to have their records deleted from the database. This information will remain dissociated from the specific information generated in the experiments.

The database will be held securely on a password-protected file server at ICO. The Principal Investigator, Dr Fernández, will designate a limited number of researchers from the UCT team to access this database.

Ethics

Informed consent: All participants taking part in the study will be properly informed orally and a written information sheet will be delivered to them. Researchers will answer all the questions that could arise during the brief session, as well as information regarding the following issues:

1. The purpose of the information to be collected, including aims, methods and implications of the research;
2. The extent to which personal data is used and accessed by the researchers (it will be made clear that all data pertaining to them is stored and handled in an anonymous manner using encrypted -not personally identifiable- codes);
3. The participant's right to access personal data and/or study data; and
4. The participant's right to withdraw from participation in the study, at any point, without consequences and without obligation of explanation or justification.

Enrolling in the study will be voluntary and signing a written informed consent will be mandatory. All original written informed consents will be stored in accordance with the Spanish legislation.

For their participation in the whole study (5 experiments in a car and 5 experiments in a room), each participant will be compensated. They will be asked to sign a compensation receipt.

Access to personal data and withdrawal from the study: It will be made clear, orally and in the information sheet, that the subjects are completely free to withdraw their records from participation in the study, regardless of having had compensation for their participation.

The consent given by participants can be withdrawn at any time, without any explanation or justification. In this case, all data pertaining to the subjects will be destroyed, both in paper and digital supports.

Human cells/tissues: Biological samples (saliva) will be collected after obtaining informed consent, in which it will be specified that these samples will be used only for the study aims, this is, the measurement of markers of tobacco-related products and other markers of exposure to aerosols from e-cigarettes, but not for the use of the cells or genetic material also contained in the saliva. The remaining saliva will be stored at the certified biobank (at ICO) and can be used for future determinations of compounds from cigarettes and e-cigarettes related to the objectives of this study.

Privacy and confidentiality: All personal information will be treated as confidential and will be stored in agreement with the current laws. The study will be conducted in accordance with the Good Clinical Practice Guidelines of the Declaration of Helsinki and the current legal regulation about the confidentiality of data in the European Union (Regulation EU 2016/679 of the European Parliament and of the Council).

Environmental protection and safety: This study will require some exposure from the participants; however, this exposure will be minimal and the participants will not be forced to be exposed if they expressed their disagreement. Similarly, the researchers will be also exposed to emissions from e-cigarettes in these confined spaces. All the researchers participating in the study will be informed and will sign a written consent for their participation.

Incidental findings: In case that while reviewing the results from the chemical analysis of nicotine metabolites in saliva any unexpected abnormality observed (what is called an "incidental finding"), the participant will be informed about it. Depending on the type of incidental finding, the participant will be contacted by mail or by phone. The participant does not have an option to decline information about an incidental finding. The costs for any care that will be needed to diagnose or treat an incidental finding would not be paid for the research study. These costs would be the responsibility of the participant.

ELIGIBILITY:
Inclusion Criteria:

For e-cigarette non-users

* Adult (18 years old and above)
* Non-e-cigarette user (never user or more than 6 months former e-cigarette user)
* Non-smoker or user of any kind of tobacco/nicotine product (never or ex-smoker for >6 months)
* Not being regularly exposed to cigarettes or e-cigarettes at home or other settings

For the e-cigarette user

* Adult (18 years old and above)
* Daily user of e-cigarettes (at least 2 months)
* Non-user of any other tobacco/nicotine products for at least 2 months

Exclusion Criteria:

For all participants:

* Pregnancy or breastfeeding
* Ongoing or recent illness (<4 weeks prior to the study)
* Acute or chronic condition or disease (diabetes, asthma, COPD, congenital heart disease, arrhythmia, hypertension or other)
* Any type of medication (<2 weeks prior to the study)

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Change in airborne nicotine concentration (mg/m3) | Pre-exposure (5 minutes*5 replications in two settings: car and room); concentration during the exposure (30 minutes*5 replications in two settings: car and room); Post-exposure (5 minutes*5 replications in two settings: car and room)
  Airborne nicotine concentration: median measurements for pre-exposure, during and post-exposure; change between pre-exposure, exposure and post-exposure periods

SECONDARY OUTCOMES:
Change in particulate matter concentration (PM2.5; mg/m3) | Pre-exposure (5 minutes*5 replications in two settings: car and room); concentration during the exposure (30 minutes*5 replications in two settings: car and room); Post-exposure (5 minutes*5 replications in two settings: car and room)
  Particulate matter concentration: median measurements for pre-exposure, during and post-exposure; change between pre-exposure, exposure and post-exposure periods
Change of in the individual exposure to tobacco related biomarkers (ng/ml) | Median concentrations at four points: before exposure, 1 minute after the exposure, 30 minutes after the end of exposure, 3 hours after the end of exposure
  Concentration of the nicotine, cotinine, TSNAs and propylene glycol in saliva samples of the participants
Changes in the irritation symptoms reported before and after exposure | Irritation symptoms at four points: before exposure, 1 minute after the exposure, 30 minutes after the end of exposure, 3 hours after the end of exposure
  Questionnaire on irritation symptoms will be administered to the participants; the change in the number of symptoms reported before and after exposure will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Esteve Fernández, Dr, Principal Investigator — Catalan Institute of Oncology (ICO) // Bellvitge Biomedical Research Institute (IDIBELL)
Locations (1):
- Catalan Institute of Oncology, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: TackSHS Project at CORDIS — https://cordis.europa.eu/project/rcn/198790/factsheet/en